CLINICAL TRIAL: NCT06367452
Title: Exploratory Pilot Study to Evaluate the Pharmacokinetic Profile of Magaldrate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tecnoquimicas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CAEP 107.001.23
Record Dates: First submitted 2024-03-20; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Alginates; Sodium Bicarbonate; magaldrate; Simethicone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taking the medication (Experimental): Participants take the standard breakfast and 30 minutes later the 10 mL suspension containing 500 mg of sodium alginate, 267 mg of sodium bicarbonate, 800 mg of magaldrate and 120 mg of simeticone
  Interventions: Drug: Sodium alginate + sodium bicarbonate + magaldrate + simeticone
- Not taking the medication (No Intervention): Participants take the standard breakfast but don't take the medication

INTERVENTIONS:
Drug: Sodium alginate + sodium bicarbonate + magaldrate + simeticone — Take an oral suspension of 10 mL 30 minutes after the ingestion of a standardized breakfast
  Other Names: Gastrofast Advance
  Arms: Taking the medication

SUMMARY:
The goal of this clinical pilot study is to evaluate the pharmacokinetic profile of magaldrate in a group of 10 healthy women, after the administration of a 10 mL drug suspension containing 500 mg of sodium alginate, 267 mg of sodium bicarbonate, 800 mg of magaldrate and 120 mg of simeticone. The main question it aims to answer is the amount of magnesium and/or aluminum, if any, absorbed into the plasma from this oral administration.

Participants will take the medication 30 minutes after a standard breakfast. Both groups of participants will take the standard meal but one group will take the medication and the other one won't.

Researchers will compare the levels of both ions in plasma in a group to see if there is any absorption, quantifying the basal plasma levels and comparing with the levels obtained after the meal and the medication, when it applies.

ELIGIBILITY:
Inclusion Criteria:

* Female participants only
* Between 18 and 55 years old
* To be available for inscription in the National Volunteers Registry for Bioequivalence studies of Brazil
* To be in good health or without any significant disease according to the responsible physician, what is stated in the protocol and the results of the laboratory tests and other tests
* To screen negativa for coronavirus (SARS-CoV-2)
* To be able to understand the nature and objective of the study, including the risks and adverse effects
* To act according to the study requirements at all times by signing the informed consent form
* The drug might bring serious risks to the fetus, so the research participant must agree to the use of a safe contraceptive method

Exclusion Criteria:

* To present flu-like symptoms that, in the medical opinion, are suspected coronavirus infection (SARS-CoV-2) within 7 days prior to the hospitalization period
* To have had direct and significant contact, in medical judgment, with individuals who tested positive for coronavirus (SARS-CoV-2) within 14 days of hospitalization
* To have a known hypersensitivity reaction to the studied medication or chemically related compounds
* Having used any medication within the 14 days prior to the hospitalization period, except contraceptives, in cases in which, based on the half-life of the medication and/or active metabolites, complete elimination can be assumed or that, at the discretion of the responsible investigator/physician, does not interfere with the pharmacokinetics or analytical stage of the study drug
* To have regularly used dietary and vitamin supplements in the 14 days before the start of the study
* To have received any dose of vaccine within the 7 days prior to the hospitalization period
* To have received, within 3 months prior to the study, treatment with any medication known to have a well-defined toxic potential in large organs
* To have participated in any experimental study or ingested any experimental medication within 6 months prior to the start of this study
* Having been hospitalized for any reason up to 8 weeks before the start of the hospitalization period of this study
* Have a history of liver disease, gastrointestinal disease, or other condition that may interfere with the absorption, distribution, metabolism, or excretion of the medication
* Have a history of kidney, respiratory, hematological, cardiac, neurological, neoplastic or psychiatric disease considered clinically significant by medical criteria
* Have a history of cardiac surgery (any type), renal surgery (renal excision or agenesis), gastrointestinal (partial or total removal of the esophagus, stomach, duodenum, jejunum, ileus, ascending colon, transverse colon, descending colon, sigmoid or rectum) and liver or pancreas surgery
* Have any current symptoms or illness, acute or chronic, under monitoring or treatment, significant at the discretion of the investigator/responsible physician
* Electrocardiographic findings not recommended at the doctor's discretion to participate in the study
* Have the results of the laboratory tests performed in the clinical evaluation of recruitment outside the values considered normal, in accordance with the reference values stipulated by the clinical analysis laboratory, unless they are considered not clinically significant by the researcher /responsible doctor
* Have laboratory test results that, according to medical evaluation, affect the safety of the research participant
* Failure to submit to coronavirus (SARS-CoV-2) testing prior to hospitalization
* Present a positive or inconclusive test for coronavirus (SARS-CoV-2) before admission
* Present a positive pregnancy test during pre-hospitalization
* Submit positive preliminary drug testing results for amphetamine/methamphetamine, opioids/morphine, marijuana/tetrahydrocannabinol, cocaine/benzoylecgonine, and/or benzodiazepine
* Being a smoker (more than 5 cigarettes/day)
* Have a history of illicit drug abuse
* Have an average alcohol intake of more than 3 doses of alcoholic beverages in a day or more than 7 doses of alcoholic beverages per week
* Having consumed alcohol and/or drugs within 48 hours before the hospitalization period
* Have the habit of drinking more than 5 cups of coffee or tea per day
* Ingest foods or drinks containing xanthines within 48 hours before hospitalization
* Eating acidic foods and/or drinks (for example, citrus fruits such as orange, tangerine, lemon, pineapple, citrus fruit juices, soft drinks, etc.) within 48 hours before the hospitalization period
* Have performed some intense physical exercise in the 48 hours before the hospitalization period
* Have unusual or restricted eating habits, at the discretion of the responsible researcher/physician
* Have donated or lost 450 mL or more of blood in the last 3 months
* Have donated or lost more than 1500 mL of blood in the last 12 months
* Having difficulty swallowing medications
* Have difficulty ingesting approximately 200 mL of water in the morning
* Presenting inability to remain awake or sitting for 1 hour or as long as necessary, at the discretion of the doctor
* Present a significant adverse event that, in the medical discretion, interferes with the safety of the participant
* Have any condition that prevents participation in the study, in the opinion of the researcher/doctor responsible

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Cmax for Aluminum | -12:00 / -06:00 / -00:10 (baseline) y 00:10 / 00:20 / 00:30 / 00:40 / 00:50 / 01:00 / 01:15 / 01:30 / 01:45 / 02:00 / 02:15 / 02:30 / 02:45 / 03:00 / 03:30 / 04:00 / 04:30 / 05:00 / 05:30 / 06:00 / 08:00 / 10:00 / 12:00 after drug administration
  To evaluate the Cmax of Aluminum to check if there is any absorption of aluminum and/or magnesium ions after oral administration of the drug in fed conditions
AUC for Aluminum | -12:00 / -06:00 / -00:10 (baseline) y 00:10 / 00:20 / 00:30 / 00:40 / 00:50 / 01:00 / 01:15 / 01:30 / 01:45 / 02:00 / 02:15 / 02:30 / 02:45 / 03:00 / 03:30 / 04:00 / 04:30 / 05:00 / 05:30 / 06:00 / 08:00 / 10:00 / 12:00 after drug administration
  To evaluate the AUC for Aluminum to check if there is any absorption of aluminum and/or magnesium ions after oral administration of the drug in fed conditions
Cmax for Magnesium | -12:00 / -06:00 / -00:10 (baseline) y 00:10 / 00:20 / 00:30 / 00:40 / 00:50 / 01:00 / 01:15 / 01:30 / 01:45 / 02:00 / 02:15 / 02:30 / 02:45 / 03:00 / 03:30 / 04:00 / 04:30 / 05:00 / 05:30 / 06:00 / 08:00 / 10:00 / 12:00 after drug administration
  To evaluate the Cmax for Magnesium to check if there is any absorption of aluminum and/or magnesium ions after oral administration of the drug in fed conditions
AUC for Magnesium | -12:00 / -06:00 / -00:10 (baseline) y 00:10 / 00:20 / 00:30 / 00:40 / 00:50 / 01:00 / 01:15 / 01:30 / 01:45 / 02:00 / 02:15 / 02:30 / 02:45 / 03:00 / 03:30 / 04:00 / 04:30 / 05:00 / 05:30 / 06:00 / 08:00 / 10:00 / 12:00 after drug administration
  To evaluate the AUC for Magnesium to check if there is any absorption of aluminum and/or magnesium ions after oral administration of the drug in fed conditions

SECONDARY OUTCOMES:
Amount of aluminum ions absorbed after drug administration vs amount provided by food | -12:00 / -06:00 / -00:10 (baseline) y 00:10 / 00:20 / 00:30 / 00:40 / 00:50 / 01:00 / 01:15 / 01:30 / 01:45 / 02:00 / 02:15 / 02:30 / 02:45 / 03:00 / 03:30 / 04:00 / 04:30 / 05:00 / 05:30 / 06:00 / 08:00 / 10:00 / 12:00 after drug administration
  To evaluate the amount of aluminum ions absorbed after drug administration compared to the amount provided by food

CONTACTS AND LOCATIONS:
Locations (1):
- CAEP, Campinas, São Paulo, Brazil

REFERENCES:
- [Derived] Burgos Castillo MJ, Cruz Palacios MJ, Iorgatchof Xavier K, Calafatti Carandina SA, Arbelaez Quintero I, do Prado Assuncao L. Evaluation of Aluminum and Magnesium Absorption Following the Oral Administration of an Antacid Suspension Containing Magaldrate in Healthy Women Under Fed Conditions. Adv Ther. 2024 Nov;41(11):4089-4097. doi: 10.1007/s12325-024-02969-9. Epub 2024 Sep 9. PMID 39249590